CLINICAL TRIAL: NCT03037424
Title: Prospective, Multi-center, Randomized, Active-control, Non-inferiority Study Comparing Fibrinogen Concentrate With Cryoprecipitate for the Treatment of Acquired Hypofibrinogenemia in Bleeding Adult Cardiac Surgical Patients
Brief Title: FIBrinogen REplenishment in Surgery
Acronym: FIBRES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Manager Anesthesia Research, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-5636-A
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Deficiency; Fibrinogen, Acquired
Keywords: Cyroprecipitate; Fibrinogen; Cardiac Surgery
MeSH Terms: interventions — cryoprecipitate coagulum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibrinogen concentrate Octafibrin (Active Comparator)
  Interventions: Drug: Octafibrin
- Cryoprecipitate (Active Comparator)
  Interventions: Drug: Cryoprecipitate

INTERVENTIONS:
Drug: Octafibrin — Octafibrin will be administered when the blood bank receives an order for fibrinogen supplementation
  Arms: Fibrinogen concentrate Octafibrin
Drug: Cryoprecipitate — Cryoprecipitate will be administered when the blood bank receives an order for fibrinogen supplementation
  Arms: Cryoprecipitate

SUMMARY:
This is a pragmatic, prospective, multi-center, randomized, active-control, single-blinded, non-inferiority phase 3 trial in adult cardiac surgical patients. Up to 12 Canadian hospitals will participate, and the trial will require up to 2 years for patient recruitment.

Twelve-hundred bleeding adult cardiac surgical patients who require fibrinogen supplementation due to acquired hypofibrinogenemia after CPB will be included. Patients will be randomized to receive equivalent doses of either fibrinogen concentrate (Octafibrin) or cryoprecipitate when the blood bank receives the first order for fibrinogen supplementation and deems it to be in accordance with accepted clinical standards. Thereafter, patients will be treated according to their assigned group each time fibrinogen supplementation is ordered during the treatment period (24 hours after termination of CPB). No other aspects of care will be modified.

The primary efficacy outcome will be the number of Allogeneic blood products (ABP) (red blood cells [RBCs], pooled or apheresis platelets, and plasma) administered during the first 24 hours after termination of CPB. Safety outcomes will be measured for the first 28 days after surgery, which is the duration of participation of each patient in the trial. Comparisons will be by intention-to-treat (ITT) (primary) and per-protocol (PP) analysis. One interim analysis will be conducted after 600 patients have been treated to determine whether the study should be terminated for safety reasons, demonstrated non-inferiority or futility reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing index cardiac surgery with CPB in whom fibrinogen supplementation is ordered in accordance with accepted clinical standards (significant hemorrhage and known or presumed hypofibrinogenemia).

Exclusion Criteria:

1. Receipt of fibrinogen rich products (fibrinogen concentrate or cryoprecipitate) within 24 hours before surgery 2. History of severe allergic reaction to cryoprecipitate or fibrinogen concentrate 3. Refusal of ABPs, fibrinogen concentrate or cryoprecipitate due to religious or other reasons 4. Fibrinogen level known to be >3.0 g/L within 30 minutes of IMP order (to eliminate the risk of raising patients' fibrinogen levels to >4.0 g/L with supplementation 5. Known pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 827 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
The primary endpoint, which is of efficacy, is the comparison of the total number of units of ABPs (RBCs, pooled or apheresis platelets, and plasma) administered during the first 24 hours after termination of CPB. | 24 hours
  The number of ABPs (red blood cells [RBCs], pooled or apheresis platelets, and plasma) administered during the first 24 hours after termination of CPB

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Karkouti, MD, Principal Investigator — University Health Network, Toronto
Locations (11):
- Canada (11):
  - Fraser University Royal Columbia, Vancouver, British Columbia
  - University of Manitoba, St Boniface General Hospital, Winnipeg, Manitoba
  - Hamilton Health Science Centre, McMaster University, Hamilton, Ontario
  - Kingston General Hsopital, Kingston, Ontario
  - London Health Science Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Tornoto General Hospital, University Health Network, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec- Université Laval, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devine C, Bartoszko J, Callum J, Karkouti K; FIBRES Study Investigators. Weight-adjusted dosing of fibrinogen concentrate and cryoprecipitate in the treatment of hypofibrinogenaemic bleeding adult cardiac surgical patients: a post hoc analysis of the Fibrinogen Replenishment in cardiac surgery randomised controlled trial. BJA Open. 2022 Jun 9;2:100016. doi: 10.1016/j.bjao.2022.100016. eCollection 2022 Jun. PMID 37588266
- [Derived] Bartoszko J, Martinez-Perez S, Callum J, Karkouti K; FIBRES Study Investigators. Impact of cardiopulmonary bypass duration on efficacy of fibrinogen replacement with cryoprecipitate compared with fibrinogen concentrate: a post hoc analysis of the Fibrinogen Replenishment in Surgery (FIBRES) randomised controlled trial. Br J Anaesth. 2022 Sep;129(3):294-307. doi: 10.1016/j.bja.2022.05.012. Epub 2022 Jun 28. PMID 35773027
- [Derived] Callum J, Farkouh ME, Scales DC, Heddle NM, Crowther M, Rao V, Hucke HP, Carroll J, Grewal D, Brar S, Bussieres J, Grocott H, Harle C, Pavenski K, Rochon A, Saha T, Shepherd L, Syed S, Tran D, Wong D, Zeller M, Karkouti K; FIBRES Research Group. Effect of Fibrinogen Concentrate vs Cryoprecipitate on Blood Component Transfusion After Cardiac Surgery: The FIBRES Randomized Clinical Trial. JAMA. 2019 Nov 26;322(20):1966-1976. doi: 10.1001/jama.2019.17312. PMID 31634905
- [Derived] Karkouti K, Callum J, Rao V, Heddle N, Farkouh ME, Crowther MA, Scales DC. Protocol for a phase III, non-inferiority, randomised comparison of a new fibrinogen concentrate versus cryoprecipitate for treating acquired hypofibrinogenaemia in bleeding cardiac surgical patients: the FIBRES trial. BMJ Open. 2018 Apr 20;8(4):e020741. doi: 10.1136/bmjopen-2017-020741. PMID 29678987